CLINICAL TRIAL: NCT02429804
Title: Combined "One Stop Shop" NaF/FDG PET/MRI Evaluation of Response to Xofigo® in mCRPC Patients: A Pilot Study
Brief Title: NaF/FDG PET/MRI in Measuring Response to Radium Ra 223 Dichloride in Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual factor
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROS0063; NCI-2015-00553 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ep 32653; 96754; PROS0063 (Other: Stanford University Hospitals and Clinics); P30CA124435 (NIH)
Record Dates: First submitted 2015-04-17; First posted 2015-04-29 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Malignant Neoplasm in the Bone; Metastatic Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (18F NaF/18F FDG PET/MRI, contrast-enhanced MRI) (Experimental): Patients receive 18F NaF and 18F FDG IV over 30 seconds-1 minute and then undergo PET/MRI and contrast-enhanced MRI after 45-60 minutes. Patients undergo imaging at baseline, after course 3 (12 weeks), and after course 6 (24 weeks) of treatment with Ra-223.
  Interventions: Procedure: Contrast-enhanced Magnetic Resonance Imaging; Drug: Fludeoxyglucose F-18; Drug: Fluorine F 18 Sodium Fluoride; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Contrast-enhanced Magnetic Resonance Imaging — Undergo contrast-enhanced MRI
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI
Drug: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Fluorine F 18 Sodium Fluoride — Given IV
  Other Names: 18 F-NaF; F-18 NaF
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot clinical trial studies combined fluorine F 18 sodium fluoride (NaF)/ fludeoxyglucose F 18 (FDG) positron emission tomography (PET) and magnetic resonance imaging (MRI) in measuring response to a drug, radium Ra 223 dichloride (Ra-223), in treating patients with prostate cancer that has not responded to hormone therapy and has spread to other parts of the body. Combining NaF/FDG in a simultaneous PET/MRI scan may help doctors accurately measure how well patients respond to treatment with radium Ra 223 dichloride.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the performance of simultaneous NaF/FDG PET/MRI for the prediction of treatment response in patients with metastatic castrate resistant prostate cancer (mCRPC).

II. Estimate the performance of simultaneous NaF/FDG PET/MRI for detection of extra-skeletal disease progression during treatment in mCRPC patients.

OUTLINE:

Patients receive 18F NaF and 18F FDG intravenously (IV) over 30 seconds-1 minute and then undergo PET/MRI and contrast-enhanced MRI after 45-60 minutes. Patients undergo imaging at baseline, after course 3 (12 weeks), and after course 6 (24 weeks) of treatment with Ra-223.

After completion of study, patients are followed up for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Diagnosed with mCRPC and painful bone metastases, referred for Xofigo (radium Ra 223 dichloride)
* Able to remain still for duration of the imaging procedure (about one hour)

Exclusion Criteria:

* Metallic implants

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Dichotomized treatment response at 24 weeks, based on technetium Tc-99m medronate (99mTc-MDP) bone scintigraphy intensity | 24 weeks
  Logistic regression of per-lesion 24-week response will be performed on percent reduction in lesion maximum standardized uptake value and percent reduction in lesion MR size. The logistic regression will include an adjustment for clustering. The receiver operating characteristic curve from the logistic regression will be graphed to give some idea of the relative sensitivity and specificity of the model.
Dichotomized treatment response at 24 weeks, based on computed tomography (CT) lesion size | 24 weeks
  Logistic regression of per-lesion 24-week response will be performed on percent reduction in lesion maximum standardized uptake value and percent reduction in lesion MR size. The logistic regression will include an adjustment for clustering. The receiver operating characteristic curve from the logistic regression will be graphed to give some idea of the relative sensitivity and specificity of the model.
Dichotomized treatment response at 24 weeks, based on alkaline phosphatase (ALP) measurements (per lesion analysis) | 24 weeks
  Logistic regression of per-lesion 24-week response will be performed on percent reduction in lesion maximum standardized uptake value and percent reduction in lesion MR size. The logistic regression will include an adjustment for clustering. The receiver operating characteristic curve from the logistic regression will be graphed to give some idea of the relative sensitivity and specificity of the model.
Percent reduction at 12 weeks in NaF/FDG PET standardized uptake value | 12 weeks
Percent reduction at 12 weeks in MRI lesion size (per lesion analysis) | 12 weeks

SECONDARY OUTCOMES:
Presence of new or regrowing extra-skeletal disease at 12 and/or 24 weeks on NaF/FDG PET/MRI that is not present on corresponding standard-of-care 99mTc-MDP bone scintigraphy and CT (per lesion analysis) | Up to 24 weeks
True status (true positive or false positive) of such lesions after 12 months of follow-up, based on all information except NaF/FDG PET/MRI (per lesion analysis) | 12 months
  The true positive fraction of progressions detected only with NaF/FDG PET/MRI will be estimated with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States